CLINICAL TRIAL: NCT02788539
Title: Reducing Disparities in the Treatment of Chronic Pain Using an Innovative mHealth Tool
Brief Title: Our Whole Lives: Online Chronic Pain Management
Acronym: OWL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Aetna, Inc. (Industry)
Responsible Party: Principal Investigator, Paula Gardiner, Assistant Professor, Boston Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: H-35182
Record Dates: First submitted 2016-05-27; First posted 2016-06-02 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; mhealth; Integrative Medicine; MBSR; Mindfulness Based Stress Reduction; Web based; Internet Based
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Science Cafe (No Intervention): One time event, Group discussion for 30 participants who are chronic pain stakeholders on pain in their community.
- Cohort 1- Pilot OWL Study (Experimental): Participants will pilot test a website- Our Whole Lives website for nine weeks in order to determine if it will help with their chronic pain management.
  Interventions: Behavioral: Our Whole Lives Website

INTERVENTIONS:
Behavioral: Our Whole Lives Website — OWL is a nine-session, web accessible, self-paced curriculum that has interactive components of self-monitoring and social support (online community).
  Arms: Cohort 1- Pilot OWL Study

SUMMARY:
This project will work to increase knowledge about the utility of a website for management of chronic pain, Our Whole Lives (OWL). It will do so by examining barriers and facilitators to patient use. In order to gather this information, the investigators will conduct a Science Cafe with 30 individuals (including participants with chronic pain, who have family members with chronic pain or are a stakeholder in the chronic pain community) to gather feedback about how to tailor the OWL website to their needs and preferences and how to improve ease of use for this tool. The investigators will also pilot two cohorts with 40 patients with chronic pain (2 groups of 20 patients) with OWL, the patient-centered, mobile health chronic pain management resource, measuring pain impact (pain severity, pain interference, physical function) and pain associated outcomes (e.g., depression, anxiety, fatigue, sleep disturbance, ability to participate in social roles and activities, pain self-efficacy, health education impact and internalized stigma related to chronic pain).

DETAILED DESCRIPTION:
During the first 4 months, conduct a science café targeting 30 individuals/families who live with chronic pain and reside in Boston's low-income, ethnically diverse neighborhoods, in order to: a) gather feedback about how to tailor the OWL curriculum based on their needs and preferences, and b) identify potential enhancements to the mobile technology to improve ease of use. For the science cafe, the investigators will use social media (facebook, twitter, listservs, etc.) to invite the community to meet for a two-hour dialog. . Each participant will be paid for attending, refreshments will be served, and a small thank you gift will be provided. Dr. Gardiner will begin the science café by giving an overview of chronic pain in the US. The moderator will ask the participants questions about how chronic pain impacts their communities and how technology might help address it.

A trained qualitative research assistant will be transcribe the science cafe and the transcripts will be analyzed using qualitative methods.

Pilot Cohort Study During the first ten months, the investigators will pilot, using pre-post measures, with 40 patients (2 groups of 20 patients) with OWL. The main outcome is pain impact (pain severity, pain interference, physical function) and pain associated outcomes (e.g., depression, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, and pain self-efficacy).

The target population includes low-income adults >18 years old who self-report: chronic musculoskeletal (extremity, joint, back, neck) pain for at least 3 months, with an average pain intensity for the previous week >4 on a 0 to 10 numerical rating scale. The investigators also require English fluency sufficient to follow instructions. Exclusion criteria include: active or planned worker's compensation, active substance abuse, psychosis, disability or personal injury claims, and known pregnancy. Participants who do not currently have access to the internet are also excluded.

The investigators will recruit patients from 14 Boston area Community Health Centers and the community of Boston Medical Center by reaching out to primary care providers for referrals. Based upon previous pilot experiences, the investigators do not anticipate any difficulty in recruiting for the pilot groups. The investigators will recruit from BMC's primary care practices and several of its 14 affiliated Community Health Centers located in Boston. Participants will receive $50 for their involvement. Based upon this initial referral, if an individual appears to be eligible for participation, he/she will be invited to meet in person with the research assistant. At this visit, eligibility is verified; the study is discussed at length with all questions answered to the participant's satisfaction; and if the patient desires, the patient enrolls by signing the informed consent. For the study, all recruitment materials will be IRB-approved prior to dissemination.

At the beginning of the study, the investigators will hold a group orientation for all 20 participants in the class on how to navigate OWL. A clinician (assisted by a RA) will demonstrate how to use the OWL system, log on, navigate through the nine sessions, complete self-assessment, set goals, and interact on the community page. Participants will have access to OWL for 9 weeks. Each week they will have access to a new content. The clinician will monitor and post questions to facilitate conversation on the community page. At the end of the 9 weeks participants will be invited back to participate in a focus group and complete 9 week follow up surveys.

ELIGIBILITY:
Inclusion Criteria:

* For Pilot Cohort Study- Chronic pain greater than or equal to 4 on a 0-10 scale for a least 12 weeks
* For Pilot Cohort Study- English comprehension sufficient to provide informed consent and understand website information.

Exclusion Criteria:

* For Pilot Cohort Study: Pregnant or planning to become pregnant in the next 3 months.
* For Pilot Cohort Study- Does not currently have access to the internet
* For Pilot Cohort Study- Begun a new pain treatment in the past month or plans to begin new pain treatments in the next 3 months.
* For Pilot Cohort Study- Does not have an internet enabled device he/she could use to access the website

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Pain Impact | 9 weeks
  a combined score of questions measuring pain severity, pain interference, and physical function. This outcome will be assessed using the PROMIS 29 scale. This information will be gathered both at baseline and in the nine week follow up survey for the two cohorts of participants pilot testing of the OWL website.

SECONDARY OUTCOMES:
Depression | 9 weeks
  These outcomes will also be assessed using the PROMIS 29 measure for the two cohorts of participants pilot testing the website at both baseline and nine weeks.
Anxiety | 9 weeks
  These outcomes will also be assessed using the PROMIS 29 measure for the two cohorts of participants pilot testing the website at both baseline and nine weeks.
Fatigue | 9 weeks
  These outcomes will also be assessed using the PROMIS 29 measure for the two cohorts of participants pilot testing the website at both baseline and nine weeks.
Sleep Disturbance | 9 weeks
  These outcomes will also be assessed using the PROMIS 29 measure for the two cohorts of participants pilot testing the website at both baseline and nine weeks.
Ability to participate in social roles and activities | 9 weeks
  These outcomes will also be assessed using the PROMIS 29 measure for the two cohorts of participants pilot testing the website at both baseline and nine weeks.

OTHER OUTCOMES:
Pain Self-Efficacy | 9 weeks
  Self-efficacy refers to capacity to persevere in the face of obstacles and adverse experiences, in this instance in the face of pain.
Perceived Stress | 9 weeks
  Perception of Stress
Internalized Stigma from Chronic Pain | 9 weeks
  Perception of stigma from chronic pain
Health Education Impact | 9 weeks
  instrument for the comprehensive evaluation of patient education programs, which can be applied across a broad range of chronic conditions

CONTACTS AND LOCATIONS:
Overall Officials: Paula Gardiner, MD,MPH, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Dresner D, Gergen Barnett K, Resnick K, Laird LD, Gardiner P. Listening to Their Words: A Qualitative Analysis of Integrative Medicine Group Visits in an Urban Underserved Medical Setting. Pain Med. 2016 Jun;17(6):1183-1191. doi: 10.1093/pm/pnw030. Epub 2016 Apr 3. PMID 27040666
- [Background] Gardiner P, Dresner D, Barnett KG, Sadikova E, Saper R. Medical group visits: a feasibility study to manage patients with chronic pain in an underserved urban clinic. Glob Adv Health Med. 2014 Jul;3(4):20-6. doi: 10.7453/gahmj.2014.011. PMID 25105072
- [Background] Saper RB, Boah AR, Keosaian J, Cerrada C, Weinberg J, Sherman KJ. Comparing Once- versus Twice-Weekly Yoga Classes for Chronic Low Back Pain in Predominantly Low Income Minorities: A Randomized Dosing Trial. Evid Based Complement Alternat Med. 2013;2013:658030. doi: 10.1155/2013/658030. Epub 2013 Jun 26. PMID 23878604
- [Background] Saper RB, Sherman KJ, Delitto A, Herman PM, Stevans J, Paris R, Keosaian JE, Cerrada CJ, Lemaster CM, Faulkner C, Breuer M, Weinberg J. Yoga vs. physical therapy vs. education for chronic low back pain in predominantly minority populations: study protocol for a randomized controlled trial. Trials. 2014 Feb 26;15:67. doi: 10.1186/1745-6215-15-67. PMID 24568299
- See also: Related Info — https://www.ourwholelives.org/